CLINICAL TRIAL: NCT06488170
Title: Patient-Reported Wellbeing Using Tildrakizumab in a Live Setting - Light Version
Brief Title: A Study to Assess Patient-Reported Wellbeing Using Tildrakizumab in a Live Setting
Status: Active, not recruiting | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: POSITIVE LIGHT
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — tildrakizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tildrakizumab: Participants who received Tildrakizumab in the frame of clinical routine for the treatment of moderate to severe plaque psoriasis in accordance with the SmPC will be observed for Week 28.
  Interventions: Drug: Tildrakizumab

INTERVENTIONS:
Drug: Tildrakizumab — As provided in real world clinical practice.
  Other Names: IL-23p19 inhibitor

SUMMARY:
The main purpose of this study to investigate the relationship between clinical symptoms and quality of life (QoL) in participants who receive Tildrakizumab in the frame of clinical routine for the treatment of moderate to severe plaque psoriasis in accordance with the summary of product characteristics (SmPC).

ELIGIBILITY:
Inclusion Criteria:

* Participant with diagnosis of moderate or severe chronic plaque PSO documented in the medical chart.
* Participant who needs systemic biologic therapy and qualifies for treatment with an IL-23p19 inhibitor. Tildrakizumab must be the anti-Il-23p19 selected therapy before including the patient in the study.
* Participant aged greater than or equal to (>=) 18 years at Inclusion.
* Written informed consent.

Exclusion Criteria:

* Participant unable or unwilling to comply with the requirements of the study.
* Participant who should not participate in the study for any reason at the discretion of the treating physician.
* Participants participating in a simultaneous clinical trial.
* Any contraindication against the use of Tildrakizumab according to the SmPC.
* Exposure to >= 3 biologics prior to inclusion.
* Participant dependent on the investigator, e.g. as employee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of participants with diagnosis of moderate-to-severe plaque psoriasis in accordance with the SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in 5-item World Health Organization Wellbeing Index (WHO-5) Score | Baseline to Week 28
  The WHO-5 is a widely used self-reported questionnaire designed to measure subjective well-being. It assesses the individual's overall psychological well-being and quality of life. The WHO-5 consists of five simple questions that ask respondents to rate their well-being over the past two weeks. The questions cover aspects such as positive mood, vitality, and general interest in life. The questionnaire is scored on a scale from 0 to 100, with higher scores indicating better well-being.

SECONDARY OUTCOMES:
Change From Baseline in Dermatology Life Quality Index (DLQI) Score | Baseline, Week 16 and 28
  DLQI is a dermatology-specific instrument used to measure the impact of skin diseases on patients' quality of life. Which assessed disease impact, monitor treatment effectiveness, guide clinical decision-making. Interpretation of Scores: 0-1: No effect on patient's life 2-5: Small effect on patient's life 6-10: Moderate effect on patient's life 11-20: Very large effect on patient's life 21-30: Extremely large effect on patient's life.
Change from Baseline in Absolute Psoriasis Area and Severity Index (PASI) Score | Baseline, Week 16 and 28
  The PASI is a measure of psoriasis and psoriatic arthritis severity that will be assessed at baseline and all follow-up visits for participants with psoriasis or psoriatic arthritis. This common clinical measure selects a representative area of psoriasis for each body region. The intensity of redness, thickness, and scaling of the psoriasis is assessed by the clinician. PASI scores range from 0 to 72, with higher scores indicating worse symptoms.
Change from Baseline in Relative PASI Score | Baseline, Week 16 and 28
  The PASI is a measure of psoriasis and psoriatic arthritis severity that will be assessed at baseline and all follow-up visits for participants with psoriasis or psoriatic arthritis. This common clinical measure selects a representative area of psoriasis for each body region. The intensity of redness, thickness, and scaling of the psoriasis is assessed by the clinician. PASI scores range from 0 to 72, with higher scores indicating worse symptoms.
Change from Baseline in Patient´s Assessment of Itch, Pain and Joint Pain as Measured by Numerical Rating Scale (NRS) | Baseline, Week 16 and 28
  NRS is the simplest and most commonly used scales to indicate the degree of pain, itch, and discomfort. The numerical scale is most commonly 0 to 10, with 0 being "no pain or Itch or discomfort" and 10 being "the worst imaginable pain or Itch or discomfort".
Number of Participants Achieving Scalp Specific Physician's Global Assessment (PGA) Score | Baseline, Week 16 and 28
  Scalp PGA assesses the overall severity of active psoriasis on the participant's scalp. Scalp lesions will be evaluated in terms of clinical signs of erythema, induration, and scaling and scored on 5-point ssPGA scale where 0=absence of disease and 4=severe disease. Higher scores indicate worsening.
Number of Participants Achieving Nail Specific PGA Score | Baseline, Week 16 and 28
  The nail specific PGA is used to evaluate the current status of a participant's nail psoriasis on a scale of 0 to 4 (clear [0], minimal [1], mild [2], moderate [3], or severe [4]).
Number of Participants Achieving Palmoplantar PGA Score | Baseline, Week 16 and 28
  The PGA is a widely used outcome measure that relies on physician visual assessment of disease severity. The PGA determines psoriasis severity at a single point in time, without taking the baseline disease condition into clear (0), almost clear (1), mild (2), moderate (3), severe (4).
Number of Participants with Psoriasis (PSO) on Family and Partners by Family PSO Questionnaire | Baseline, Week 16 and 28
  PSO is a self-administered questionnaire designed to address impact of PSO on family and partners by Family PSO questionnaire. Family PSO is a self-administrated questionnaire to assess the burden on partners of patients with psoriasis. The questionnaire has 15 items divided into five factors: (1) perceived strain by social reactions to the partner's psoriasis; (2) strain caused by cleaning; (3) acute emotional strain attributed directly to the psoriasis; (4) restrictions of social life; and (5) general emotional strain. The items are scaled in a 5-point Likert format: 0='not true', 1='somewhat true', 2='moderately true', 3='quite true', 4='very true', with the supplementary option 'does not apply to me'.
Number of Participants with Psoriasis Treatment on Physician's Satisfaction | Baseline, Week 28
Hospital Anxiety and Depression Scales (HADS) Questionnaire | Baseline, Week 16 and 28
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). A score between 0 and 7 is 'normal', between 8 and 10 shows "light" level, between 11 and 14 "moderate" level, and between 15 and 21 "severe" level of anxiety/depression.
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Baseline, Week 16 and 28
  FACIT-F is a questionnaire-based tool (FACIT-F, Vision 4) used to measure fatigue in patients. It consists of multiple items, each focusing on a different aspect of fatigue. The items are typically rated on a scale from 0 to 4, with 0 representing "not at all" and 4 representing "very much". Example items include: "I feel tired" or "I'm too tired to working". Higher scores indicate less fatigue.
Correlations Between the Aforementioned Parameters, in Particular WHO-5 and HADS | Baseline, Week 16 and 28
  To determine the correlation between the aforementioned parameters, in particular WHO-5 and HADS. Correlations between parameters are tested by the non-parametric Spearman test. In case of significant correlations, and if the nature of the data allows it, the conduct of more advanced regression analyses is permissible.
Correlations Between the Aforementioned Parameters, in Particular WHO-5 and FACIT-F | Baseline, Week 16 and 28
  To determine the correlation between the aforementioned parameters, in particular WHO-5 and FACIT-F. Correlations between parameters are tested by the non-parametric Spearman test. In case of significant correlations, and if the nature of the data allows it, the conduct of more advanced regression analyses is permissible.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, S.A.
Locations (7):
- Czechia (7):
  - University Hospital Ostrava, Ostrava
  - Fakultní nemocnice Plzeň, with its registred seat at Edvarda Beneše, Pilsen
  - University Hospital Kralovske Vinohrady, Prague
  - University Hospital in Motol, Prague
  - General university hospital Prague, Prague
  - University Hospital Bulovka, Prague
  - Masarykova hospital Ústí nad Labem, Ústí nad Labem

IPD SHARING:
Plan to Share IPD: No